CLINICAL TRIAL: NCT05204199
Title: Towards Individualization of Bladder Cancer Therapy: the Role of Microbiome in BCG Responsiveness Prediction
Brief Title: Role of Microbiome in BCG Responsiveness Prediction
Acronym: SILENTEMPIRE
Status: Recruiting | Type: Observational
Sponsor: Cédric Poyet (Other)
Collaborators: Krebsliga Schweiz (Unknown)
Responsible Party: Sponsor-Investigator, Cédric Poyet, Principal Investigator, University of Zurich
Organization: University of Zurich (Other)
Other Study IDs: 2021-01783
Record Dates: First submitted 2021-12-29; First posted 2022-01-24 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Microbiome; Bladder Cancer
Keywords: BCG
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Bladder tissue samples, fecal samples, Instrumented urine samples, blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group A: Patients without a urological or gastrointestinal malignancy undergoing non-oncological bladder surgery or transurethral resection of the prostate (TUR-P)
- Group B: Low Risk NMIBC (primary, solitary, Ta / low grad < 3cm, no carcinoma in situ (CIS))
- Group C: NMIBC patients, BCG candidates, assessed as intermediate (between the category of low- and high risk) or high risk (T1 or high grade or CIS or multiple, recurrent and large (> 3 cm) Ta/ low grade tumours).

SUMMARY:
Our primary aim is to investigate the use of microbial profile from the bladder and the feces of NMIBC patients as a predicting tool for therapy response prior to BCG administration.

Our second aim is to collect additional samples (blood, instrumented urine, bladder tissue, feces) to establish a local biobank for future microbiome projects.

DETAILED DESCRIPTION:
The microbiome, defined as a characteristic microbial community occupying a reasonably well-defined environment (e.g. gut microbiome), has been increasingly linked with different medical conditions and also with cancer. While there have been numerous investigations into the gut bacterial ecosystem, scientists have started to pay attention to the microbiome of the bladder only recently. Results from newest investigations support the understanding that the bladder possesses its own microbiome and it is not germ-free. Studying the relationship between bladder cancer and bladder and gut microbiome may lead to new insights which can be used to predict tumor behavior and/or response to therapy.

With this project, we aim to investigate the use of microbial fingerprint from the bladder and from the feces of bladder cancer patients in predicting therapy response prior to administration of Bacillus Calmette-Guerin or BCG. BCG causes the body's own immune system to attack the bladder cancer cells. It is applied directly into the bladder to prevent the cancer from growing and from regrowing. However, in around 40% of patients this treatment is not successful, BCG should be avoided, and other therapy strategies should be chosen. Unfortunately, there is no test available yet, which help to select patients who will benefit from the therapy before the therapy is started.

In this project we intend to determine the microbial fingerprint and to analyze if this fingerprint can be used as a selection tool. This tool may enable as us in the future to avoid application of BCG therapy for patient with a high risk of therapy failure and save time to start alternative therapy options and hopefully avoid tumor progression. Our second aim is to collect additional samples (blood, instrumented urine, bladder tissue, feces) to establish a local biobank for future microbiome projects.

ELIGIBILITY:
Inclusion Criteria

* Signed informed consent
* Ability to understand and follow study procedures and understand informed consent
* age 18 - 90 years

Exclusion Criteria

* Antibiotic treatment within the last month
* Immuno-/chemotherapy within the past 6 months
* Immunosuppressive therapy
* Major medical, neoplastic (with the exception of skin cancer), surgical or psychiatric condition requiring ongoing management. Minor, well-controlled conditions, such as medically controlled arterial hypertension or occupational asthma, may be present.
* Additional major diagnosis known to affect the gut or bladder microbiota (e. g. liver cirrhosis, systemic sclerosis, inflammatory bowel disease, inflammatory bowel syndrome, celiac disease, neuropathic bladder)
* Major past intestinal surgery, especially in small intestine or colon. Cholecystectomy, appendectomy, past perianal surgery or past hernia repair may be present.
* Major gastrointestinal symptoms (diarrhoea, constipation, abdominal pain, vomiting, unexplained weight loss, rectal bleeding or blood in the stool)
* Bladder augmentation surgery.
* Indwelling urinary catheter

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Group A: Patients without a urological or gastrointestinal malignancy undergoing non-oncological bladder surgery or transurethral resection of the prostate (TUR-P) fulfilling the following criteria. At the time of study inclusion, no urological symptoms or relevant urological disease (Unclear Macrohematuria, Cystolithiasis, prostate Cancer )
  Group B: Low Risk NMIBC (primary, solitary, Ta / low grad < 3cm, no carcinoma in situ (CIS)).
  Group C: NMIBC patients, BCG candidates, assessed as intermediate (between the category of low- and high risk) or high risk (T1 or high grade or CIS or multiple, recurrent and large (> 3 cm) Ta/ low grade tumours).
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-02-22 (Actual); Primary Completion 2025-10-20 (Estimated); Study Completion 2025-10-20 (Estimated)

PRIMARY OUTCOMES:
Difference in microbial Profile | 1 year
  use of microbial profile from the bladder and the feces of NMIBC patients as a potential binary classification system, to substratify BCG-candidates into "anticipated BCG-responder (aBCGr)" and "anticipated BCG-non-responder (aBCGnr)" groups in predicting therapy response prior to BCG administration.

SECONDARY OUTCOMES:
Biobank | 1 year
  collect additional samples (blood, instrumented urine, bladder tissue, feces) to establish a local biobank for future microbiome projects

CONTACTS AND LOCATIONS:
Overall Officials: Cédric Poyed, MD, Principal Investigator — University Hospital Zurich, Departement of Urology
Locations (5):
- Switzerland (5):
  - Kantonsspital Baden, Baden, Canton of Aargau
  - Spitalzentrum Biel, Biel/Bienne, Canton of Bern
  - Kantonsspital St. Gallen, Sankt Gallen, Canton of St. Gallen
  - Kantonsspital Winterthur, Winterthur, Canton of Zurich
  - University Hospital Zürich, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bieri U, Scharl M, Sigg S, Szczerba BM, Morsy Y, Ruschoff JH, Schraml PH, Krauthammer M, Hefermehl LJ, Eberli D, Poyet C. Prospective observational study of the role of the microbiome in BCG responsiveness prediction (SILENT-EMPIRE): a study protocol. BMJ Open. 2022 Apr 18;12(4):e061421. doi: 10.1136/bmjopen-2022-061421. PMID 35437256